CLINICAL TRIAL: NCT02833896
Title: Endometrial Cancer: Evaluation of Genetic Imbalances in the Carcinogenesis Process
Brief Title: Endometrial Cancer and Array CGH
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA11019
Record Dates: First submitted 2016-07-04; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Cancer of the Endometrium
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- endometrial cancer
  Interventions: Genetic: surgery
- Control
  Interventions: Genetic: surgery

INTERVENTIONS:
Genetic: surgery

SUMMARY:
Medical context:

Several molecular studies showed chromosomal alterations in patients with endometrial cancer, with gains in 1q, 19p, 19q, 8q, 10q and 10p and loss of 4q, 16q and 18q. Several genes of interest have been dentified (P53, PTEN, PIK3CA, ß-catenin, K-ras ...). It is thus conceivable that like that enable genomic tools used in breast cancer today (Oncotype DX, MammaPrint), correlation between the tumor profile and life project in the case of cancer the endometrium could be done. A study is already underway at the Reims University Hospital with funding from the League against cancer and AOL in 2010 CHU Reims. It should identify the specific alterations of nosologic continuum of pathology and characterize areas of interest on the genome. To date, 39 patients with endometrial cancer and 15 patients with endometrial hyperplasia (patients 'cases') were included in the study. For this study, 10 patients exhibiting neither cancer nor endometrial hyperplasia were also included. Samples of these 10 patients 'witnesses' were pooled to serve as a reference for analyzing patients 'cases'.

objectives: In continuation of the study began in November 2009, refine the study of genomic imbalances highlighted hyperplasia and endometrial cancer by studying the in correlation between genomics and proteomics by immunohistochemical studies and analyzing the microsatellite instability.

To study the prognostic role of genetic factors in patients carriers of a disease endometrial (cancer or hyperplasia).

Material and methods :

Experimental Design: Cross-sectional study in inclusion prospective multi-center followed by a cohort study of patients 'cases'.

Population / patients: in total, it is planned to include 72 patients with hyperplasia or endometrial cancer (22 patients included in the pre-study part funded by the League against cancer 50 patients included in the scope of the study funded by the 2010 AOL Chu Reims).

Plan of investigation: the study includes two phases:

Sectional study:

The inclusion of 10 patients "witnesses" has already been completed in the first project.

During the consultation in the obstetrics and gynecology department of the Reims University Hospital and the surgical department of the institute Jean Godinot, terms and objectives of the study have been and will be presented to patients where cancer or hyperplasia endometrial was diagnosed by achieving endometrial biopsy.

If the patient agrees to participate in the study, the management of its pathology (hysterectomy, hysteroscopy and curettage resection) will not be changed.

The samples taken during the surgery were analyzed and will be as provided in the first research project. Tumor karyotype, DNA extraction are performed on each sample fresh. A comparative genomic hybridization is conducted using the DNAs thus obtained.

Additional analyzes (immunohistochemistry and analysis of microsatellite instability) will be performed on all samples already obtained and on future withdrawals.

ELIGIBILITY:
Inclusion Criteria:

* Having a pathological diagnosis of hyperplasia or endometrial cancer
* consent to participation in the study

Exclusion Criteria:

* Not affiliated to a social security scheme

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with cancer or hyperplasia endometrial
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2010-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
quantitative analysis of Ki67 by immunohistochemistry analysis | up to 1 year
quantitative analysis of P53 by immunohistochemistry analysis | up to 1 year
quantitative analysis of HER2 by immunohistochemistry analysis | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France